CLINICAL TRIAL: NCT00002259
Title: Phase II Study of Intravenous Novantrone(R) in the Treatment of AIDS Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lederle Laboratories (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 055B; 3-102
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-08

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Mitoxantrone; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Mitoxantrone

INTERVENTIONS:
Drug: Mitoxantrone hydrochloride

SUMMARY:
To study the toxicity and efficacy of IV mitoxantrone hydrochloride (Novantrone) in AIDS-related Kaposi's sarcoma.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Biopsy proven Kaposi's sarcoma in advanced stages.
* Positive HIV antibody, HIV culture or antigen capture or T4 cells < 500 in a patient with AIDS risk factor.
* Informed consent and availability for follow-up.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Uncontrolled opportunistic infection.
* Any medical, surgical or psychiatric condition which would constitute a contraindication to the use of mitoxantrone.

Concurrent Medication:

Excluded:

* Zidovudine (AZT).

Patients with the following are excluded:

* Uncontrolled opportunistic infection.
* Unable to give informed consent.
* Any medical, surgical or psychiatric condition which would constitute a contraindication to the use of mitoxantrone.

Prior Medication:

Excluded:

* More than one form of chemotherapy regimen.
* Doxorubicin therapy > 300 mg/m2.

Prior Treatment:

Excluded:

* Previous therapy consisting of more than one modality of therapy (e.g., chemotherapy plus radiotherapy or more than one form of chemotherapy regimen.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Luke's - Roosevelt Hosp Ctr, New York, New York, United States